CLINICAL TRIAL: NCT03371043
Title: Outpatient Use of Analgesics in Children and Adolescents in France
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 15FKU-Analgesic
Record Dates: First submitted 2016-09-07; First posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Outpatient Use of Analgesics in Children and Adolescents
Keywords: analgesics; opioids; outpatient drug use; pediatrics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- users of analgesic medications: Children and adolescents who are users of analgesic medications, 2012 to 2015
  Interventions: Other: users of analgesic medications

INTERVENTIONS:
Other: users of analgesic medications — Children and adolescents who are users of analgesic medications, 2012 to 2015

SUMMARY:
outpatient use of analgesics in children and adolescents in France from 2012 to 2015

DETAILED DESCRIPTION:
To describe the outpatient use of analgesics in children and adolescents in France from 2012 to 2015

ELIGIBILITY:
Inclusion Criteria:

* all children and adolescents (0-17 years)
* registered in the French Health Insurance Database from 2012-2015

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and adolesents who are users of analgesic medications, 2012 to 2015
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Analgesic and anti-migraine drugs with a specific focus on opioids | 4 years
  Quantification of the use of analgesics and changes over time

SECONDARY OUTCOMES:
Co-analgesic drugs (antidepressants and anticonvulsants) for pain management | 4 years
  Use of co-analgesics. children and adolescents with epilepsy or a psychiatric disorder will be excluded from the main analysis in order to approximate as much as possible the use of these drugs for pain management Acute or chronic use Geographical distribution of prescribers For co-analgesics specifically: description of analgesic drugs used concomitantly.
  Assessment of off-label use of analgesics by comparing descriptive usage data and regulatory marketing authorization conditions: for each analgesic; age of use and use of codeine in off-label indications will be assessed
Description of outpatient use of opioid analgesics over time in children with malignant disease | 4 years
  Types of specific molecule and drug combinations: Assessment of these parameters will concern two distinct periods of time: ≤1 year after the diagnosis of cancer disease and >1 year after diagnosis. The diagnosis date will either the date of the first hospitalization for cancer or the date of full expenses coverage by the health insurance system for cancer disease, whichever comes first.
  Profile of prescribers: hospital or private practice Profile of patients: age groups (0-23 months, 2-5 years, 6-11 years, 12-17 years) Acute or chronic use. Chronic use will be defined by at least 3 dispensations of the same analgesic drug (ATC code 5th level) in a period of 12 months.
Evaluation of the dispensing without medical prescription of analgesics in children and adolescents. | 4 years
  Proportion of analgesics' dispensations without medical prescription presented by age and gender

CONTACTS AND LOCATIONS:
Overall Officials: Florentia Kaguelidou, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Robert Debré, APHP, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided